CLINICAL TRIAL: NCT07397663
Title: Prediction of Intradialytic Hypotension at the Initiation of Continuous Venovenous Hemodiafiltration Using Multimodal Ultrasonographic and Hemodynamic Parameters in Intensive Care Unit Patients
Brief Title: Ultrasound-Based Prediction of Hemodynamic Instability During CVVHDF Initiation
Acronym: US-CVVHDF
Status: Not yet recruiting | Type: Observational
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Musa Harun UÇAR, Specialist physician, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: registration pending
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Renal Failure , Chronic; Intradialytic Hypotension; Critical Illness
Keywords: Intradialytic Hypotension; LVOT VTI; CVVHD; Renal Resistive Index; Echocardiography; VExUS
MeSH Terms: conditions — Renal Insufficiency, Chronic; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational study aims to evaluate the ability of transthoracic echocardiographic and bedside ultrasonographic parameters to predict intradialytic hypotension and hemodynamic instability at the initiation of continuous venovenous hemodiafiltration (CVVHDF) in adult intensive care unit patients.

DETAILED DESCRIPTION:
In critically ill patients requiring renal replacement therapy, continuous venovenous hemodiafiltration (CVVHDF) is frequently preferred due to better hemodynamic tolerance. However, initiation of CVVHDF may still lead to unpredictable intradialytic hypotension, fluid requirement, or vasopressor/inotrope support.

Bedside transthoracic echocardiography and ultrasonography provide non-invasive assessment of cardiac function, preload responsiveness, and venous congestion. Parameters such as left ventricular outflow tract velocity time integral (LVOT VTI), mitral annular plane systolic excursion (MAPSE), tricuspid annular plane systolic excursion (TAPSE), pulse pressure variation (PPV), renal resistive index (RRI), inferior vena cava (IVC) diameter, and venous excess ultrasound score (VExUS) may help predict hemodynamic tolerance to dialysis.

This study aims to evaluate the predictive value of these multimodal ultrasonographic and hemodynamic parameters for intradialytic hypotension and hemodynamic support requirement during the first 60 minutes of CVVHDF initiation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) admitted to the intensive care unit
* Indication for continuous venovenous hemodiafiltration
* Adequate transthoracic echocardiographic image quality
* Written informed consent obtained from legal representatives

Exclusion Criteria:

* Acute coronary syndrome
* Severe valvular heart disease or pericardial effusion
* Significant arrhythmias interfering with Doppler measurements
* Presence of pacemaker, ICD, or ventricular assist device
* Poor echocardiographic imaging window
* Life expectancy less than 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (aged 18 years and older) admitted to the intensive care unit of a tertiary care academic hospital who have a clinical indication for continuous venovenous hemodiafiltration (CVVHDF).
  All participants are critically ill and require renal replacement therapy as part of standard clinical care. Transthoracic echocardiography and bedside ultrasonographic and hemodynamic assessments are performed as part of routine intensive care evaluation and are recorded for observational purposes only.
  No healthy volunteers are included in this study. Written informed consent is obtained from the patients' legal representatives prior to study inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2027-02-10 (Estimated); Study Completion 2027-02-10 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic Instability During CVVHDF Initiation | First 60 minutes after CVVHDF initiation
  Occurrence of hypotension (mean arterial pressure <65 mmHg), requirement for fluid bolus (≥500 mL), or initiation/increase of vasopressor or inotrope support within the first 60 minutes after CVVHDF initiation.

SECONDARY OUTCOMES:
LVOT Velocity Time Integral | Before CVVHDF initiation
  Measurement of left ventricular outflow tract velocity time integral obtained by transthoracic echocardiography before dialysis initiation.
Mitral Annular Plane Systolic Excursion (MAPSE) | Before CVVHDF initiation
  Measurement of mitral annular plane systolic excursion obtained by M-mode transthoracic echocardiography in the apical four-chamber view to assess left ventricular longitudinal systolic function prior to CVVHDF initiation.
Tricuspid Annular Plane Systolic Excursion (TAPSE) | Before CVVHDF initiation
  Measurement of tricuspid annular plane systolic excursion obtained by M-mode transthoracic echocardiography in the apical four-chamber view to evaluate right ventricular systolic function prior to CVVHDF initiation.
Pulse Pressure Variation (PPV) | Before CVVHDF initiation
  Calculation of pulse pressure variation derived from invasive arterial blood pressure waveform analysis in mechanically ventilated patients to assess dynamic preload responsiveness prior to CVVHDF initiation.
Renal Resistive Index (RRI) | Before CVVHDF initiation
  Measurement of renal resistive index obtained by pulsed-wave Doppler ultrasonography of segmental or interlobar renal arteries to evaluate intrarenal vascular resistance and renal perfusion prior to CVVHDF initiation.
Inferior Vena Cava Diameter | Before CVVHDF initiation
  Ultrasonographic measurement of inferior vena cava diameter obtained from the subcostal long-axis view to assess intravascular volume status prior to CVVHDF initiation.
Venous Excess Ultrasound Score (VExUS) | Before CVVHDF initiation
  Assessment of systemic venous congestion using the Venous Excess Ultrasound Score (VExUS), incorporating inferior vena cava diameter and Doppler flow patterns of hepatic, portal, and renal veins prior to CVVHDF initiation.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Cheong I. Unconventional Echocardiographic Techniques for LVOT VTI Measurement in Critical Care Settings. J Clin Ultrasound. 2025 Jul-Aug;53(6):1418-1424. doi: 10.1002/jcu.24007. Epub 2025 Apr 12. PMID 40219729
- [Background] Assavapokee T, Rola P, Assavapokee N, Koratala A. Decoding VExUS: a practical guide for excelling in point-of-care ultrasound assessment of venous congestion. Ultrasound J. 2024 Nov 19;16(1):48. doi: 10.1186/s13089-024-00396-z. PMID 39560910
- [Background] Monnet X, Shi R, Teboul JL. Prediction of fluid responsiveness. What's new? Ann Intensive Care. 2022 May 28;12(1):46. doi: 10.1186/s13613-022-01022-8. PMID 35633423
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/39560910/
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC5668149/